CLINICAL TRIAL: NCT05937321
Title: NIDDK Share Plus: Continuous Glucose Monitoring with Data Sharing in Older Adults with T1D and Their Care Partners
Brief Title: National Institute of Diabetes and Digestive Kidney Diseases* Share Plus: Continuous Glucose Monitoring with Data Sharing in Older Adults with Type 1 Diabetes* and Their Care Partners to Improve Time in Range and Reduce Diabetes Distress.
Acronym: NIDDK T1D
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Nancy Ann Allen, Associate Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00160673
Record Dates: First submitted 2023-06-21; First posted 2023-07-10 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: T1D; diabetes; cgm; telehealth; care partner; data sharing; diabetes education; older adult
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — Methods; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group- Virtual with Dyad Follow + Share plus (Experimental): The Share plus intervention is a behavioral intervention administered by a certified diabetes education and care specialist (CDCES) using telehealth. Share plus consists of three educational sessions to facilitate dyads' success in data sharing glucose levels. The Share plus intervention has five major components that are delivered using techniques of motivational interviewing: 1) shared appraisal, 2) communication strategies, 3) problem-solving strategies, 4) action planning and, 5) re-evaluating, practicing, and advancing.
  Interventions: Behavioral: Share plus intervention
- Control Group- Virtual with Dyad Follow + Diabetes Self-Management Education (Active Comparator): Participants will receive diabetes self-management education using the Association of Diabetes Care and Education Specialists 7 education curriculum (ADCES7).
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: Share plus intervention — Participants will receive the Share plus intervention:
  * Set up Follow app
  * Start Share plus intervention
  * Communication and problem-solving strategies
  * Detailed action plan including glucose targets
  * Review communication and problems
  * New communication content
  * Revise action plan as needed for communication and problem-solving hypo- and hyperglycemia,
  * Dyadic glucose pattern management training using Clarity, set automatic Clarity downloads
  * Dyad set goals for regular times to discuss glucose trends and problem-solving
  * Dyadic review of glucose targets after an in-depth analysis of CGM data and dyadic treatment strategies to improve glucose TIR
  Arms: Intervention Group- Virtual with Dyad Follow + Share plus
Behavioral: Control group — Diabetes self-management education materials
  Arms: Control Group- Virtual with Dyad Follow + Diabetes Self-Management Education

SUMMARY:
The purpose of this study is to test the Share plus intervention aimed at improving the use of data sharing between people with diabetes and their care partners in order to maximize the benefits of continuous glucose monitoring.

Hypothesis: Compared to the control group, persons with diabetes enrolled in the Share plus intervention group will experience clinically significant improvements in time-in-range (TIR) (>5%) at 12- and 24-weeks into the study, and improvement on diabetes distress. Care partners enrolled in the Share plus intervention group will experience lower diabetes distress at 12- and 24-weeks into the study.

DETAILED DESCRIPTION:
Older adults with type 1 diabetes (T1D) have an increased risk of hypoglycemia and hyperglycemia that can result in grave health consequences, such as seizures, falls, and myocardial infarctions. Care partners (e.g., spouses, friends) regularly become part of the diabetes care team to assist in self-management as a person with diabetes ages. A technological advancement that is available to people with diabetes and their care partners to address harmful hypoglycemia and hyperglycemia is to use continuous glucose monitoring (CGM), with a data-sharing app that allows the older adult with T1D and their care partner (dyad) to see glucose data on their smart-phones and to receive an alert before hypoglycemia or hyperglycemia occurs. Our long-term goal is to leverage the full potential of technology and care partner interventions to optimize the support that care partners can provide for effective glucose management in older adults with T1D. Our overall objective is to test an intervention, called Share plus, aimed at improving the use of data sharing between persons with diabetes and their care partners in order to maximize the benefits of CGM. The Share plus intervention provides instruction to current CGM users about how to set up the data sharing app, dyadic communication and problem solving, and how to establish a data-sharing action plan for older adults with T1D and their care partners.

Our central hypothesis is that Share plus will result in increased time-in-range and decreased diabetes distress for both persons with diabetes (PWD) and their care partners (CPs) compared to the control group. The rationale for this pilot study is that demonstrating the efficacy of Share plus will provide new opportunities for a clinically useful approach to increase time in glucose range and decrease diabetes distress among older adults with T1D and their care partners. The central hypothesis will be tested by pursuing three specific aims: 1) evaluate feasibility, usability, and acceptability of the Share plus intervention compared to the control group receiving data sharing with diabetes self-management education, 2) evaluate the effect of Share plus intervention on time-in-range and Diabetes Distress, and 3) explore the differences between groups in PWD and CP dyadic appraisal and coping, quality of life, diabetes self-care and care partner burden. To test our central hypothesis, we will conduct a pilot randomized 1:1 control trial in older adults with T1D already using CGM (N=80 dyads) in a telehealth format where the intervention group will receive data sharing and Share plus and the control group will receive diabetes self-management education and assistance setting up the data sharing app. The trial will include a 12-week active intervention to determine a change in primary outcomes and a 12-week observation-only phase to determine maintenance of changes. The research proposed in this application is innovative because it provides a needed and substantive departure from the status quo by bringing a dyadic perspective of T1D management using data-sharing technology.

ELIGIBILITY:
Inclusion Criteria for PWD:

* 60 + years of age
* Type 1 Diabetes Diagnosis
* HbA1c no greater than 11.0%
* Currently using continuous glucose monitoring
* Able to manage diabetes with respect to insulin administration and glucose monitoring (which may include assistance from a care partner

Inclusion Criteria for CP:

* ≥18 years of age
* Participant understands the study protocol and agrees to comply with it

Exclusion Criteria for PWD:

* Life expectancy estimated at < 1 year
* Extreme visual or hearing impairment that would hinder the ability to use CGM
* Stage 4 or 5 renal disease or most recent Glomerular filtration rate (GFR) <30 ml/min/m2 from a local lab within the past six months
* The presence of a significant medical or psychiatric condition or use of a medication that in the investigator's judgment may affect the completion of any aspect of the protocol.
* Clinical diagnosis of moderate or severe dementia
* Inpatient psychiatric treatment in the past six months
* Participation in an intervention study in the past six weeks
* Montreal Cognitive Assessment Score < 19

Exclusion criteria for CP:

* Cognitive impairment or dementia
* Medical condition that will make it inappropriate or unsafe to fulfill the role of a CP

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-11-02 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Time in Range | Change from 12 weeks to 24 weeks
  Time in Range equals 70-180 mg/dl, collected from Clarity reports- 14 days at each timepoint; glycemic metrics: collect from Clarity report - 14 days including hypoglycemic range (less than 60 mg/dl), hyperglycemic range (181-249 and greater than 250 mg/dl), and glycemic variability coefficient value; Hemoglobin A1C (A1C): Collected via home A1c test kits, provided and processed by University of Minnesota Advanced Research and Diagnostic Laboratory.

SECONDARY OUTCOMES:
Diabetes Distress for Adults with Type 1 Diabetes | Change 12 weeks to 24 weeks
  28 items. Minimum score is 0 and maximum score is 28. A higher score indicates a worse outcome.
Diabetes Distress Scale for Partners of Adults with Type 1 Diabetes | Change 12 weeks to 24 weeks
  21 items. Minimum score is 0 and maximum score is 21. A higher score indicates a worse outcome.

OTHER OUTCOMES:
Diabetes Appraisal | Change 12 weeks to 24 weeks
  1 item. Minimum score is 1 and maximum score is 3. The lower the score the worse the outcome.
Supportive and Unsupportive Behaviors | Change 12 weeks to 24 weeks
  15 items. The minimum score is 15 and the maximum score is 75. A lower score on the Emotional Support, Instrument Support and Collaboration subscales indicate a worse outcome. A higher score on the Unsupportive/controlling scale indicates a worse outcome.
Quality of Relationships Inventory | Change 12 weeks to 24 weeks
  24 items. Minimum score is 24 and maximum score is 120. The lower the score the worse the outcome.
Care Partner Burden | Change 12 weeks to 24 weeks
  1 item. Minimum score is 1 and maximum score is 5.
Diabetes Self-Care Inventory Revised | Change 12 weeks to 24 weeks
  15 Items. Minimum score is 15 and maximum score is 75. The lower the score the worse the outcomes.
World Health Organisation-Five Well-Being Index | Change 12 weeks to 24 weeks
  The minimum score is 0 and the maximum score is 100. Lower scores indicate worse well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy A Allen, PhD, Principal Investigator — University of Utah College of Nursing
Locations (1):
- University of Utah College of Nursing, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Allen NA, Berg CA, Iacob E, Gonzales BR, Butner JE, Litchman ML. Examining Share plus-A Continuous Glucose Monitoring Plus Data-Sharing Intervention in Older Adults and Their Care Partners: Protocol for a Randomized Control Study. JMIR Res Protoc. 2024 Dec 16;13:e60004. doi: 10.2196/60004. PMID 39680874